CLINICAL TRIAL: NCT07177170
Title: Optimizing Cervical Cancer Screening Strategies With HPV Testing Among Women Living With HIV in Cameroon: Feasibility, Acceptability, and Impact of a Single-visit Test and Treat Approach in a Hospital Center With an HPV Testing Platform
Brief Title: Impact of a Single Versus Multiple Visits on the Cervical Cancer Screening Completeness, Feasibility and Acceptability Among Women Living With HIV in Cameroon
Acronym: OptiTri_GC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other); Centre Pasteur du Cameroun (Other); Centre Hospitalier Simone VEIL de BEAUVAIS (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Queen Mary University of London (Other); Hôpitaux Universitaire de Genève (Unknown); International Agency for Research on Cancer (Other); Programme PACCI, Abidjan, Côte d'Ivoire (Unknown); RSD Institute, Cameroon (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: IRD_2024_CEPED_OptiTri_GC; 22SANIC204 (Other Grant/Funding Number: Initiative); ANRS-0467 (Other Grant/Funding Number: ANRS-MIE)
Record Dates: First submitted 2025-08-22; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer Screening; HIV
Keywords: cervical cancer; screening; HIV; differentiated prestation; implementation; resource-limited setting; thermal ablation; HPV test
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design ("before - after") combined with a case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single visit (Active Comparator): All women will be screened using a single-visit approach
  Interventions: Other: Single visit
- Differentiated prestation (Experimental): A more flexible screening approach will be offered based on the participants preference. After counseling (following the decision aid approach), participants may decide to performed the screening in two visits.
  Interventions: Other: Differentiated screening delivery

INTERVENTIONS:
Other: Differentiated screening delivery — More flexibility in the screening delivery will be offered. A decision aid process will be implemented to help the participants deciding between the two options.
  Arms: Differentiated prestation
Other: Single visit — All the steps of the screening (using HPV test) and of the treatment will be performed in a single visit (when possible).
  Arms: Single visit

SUMMARY:
Context. Cervical cancer (CC) is a leading cause of death among women living with HIV (WLHIV) in resource-limited settings. Yet, effective methods for screening and preventing CC are available. The recommanded approach for CC screening is based on multiple steps, including initial test to detect human papillomavirus (HPV) infection, visual inspection to identify women with HPV at risk for precancerous lesion and treatment when required.

Dropout may occur at these different steps, compromising the success of the CC elimination strategy. Performing the all screening and treatment sequence in a single visit has been recommanded based on the results of a large South African trial. Yet, in many contexts, including those with limited resources, the screening and treatment activities are performed in multiple visites for logistical reasons, resulting in many dropouts. Strategies based on the differentiated prestation approaches, which propose a simplified management centered on the patients preferences, could guide the adaptation of the single-visit approach to account for contextual constraints while maintaining high effectiveness.

The OptiTri-GC study aims to design and assess the impact of a differentiated CC screen and treat strategy in a district hospital; It will assess both its implementation and its effectiveness based on the completeness at each stage of the screening cascade. In addition, it will also include three sub-studies designed to evaluate :

* The performance of urinary HPV testing.
* The performance of different methods to identify women requiring a treatment.
* The risk of post-treatment cervical disease.

This study has two periods. During the first period, a single visit approach will be used while differentiated approach will be prepared using participatory research. During the second period, the differentiated approach will be implemented. The screening overall completeness will be compared between the two periods to assess the differentiated approach effectiveness.

The study will also assess the implementation of each screening strategy in terms of :

* Success through the measure of fidelity, reach and completeness
* Identification of adaptation, barriers and facilitating/leverage factors
* Perception, feasibility and acceptability of the screening strategies (by patients and health care workers) It will assess the participants' stress levels during the screening process and to identify potential psychosocial support strategies and document the experience of WLHIV and health workers during the screening process and the post-treatment follow-up.

Other study objectives include :

* To assess the performance of different methods to identify women requiring a treatment
* To assess the performance of HPV testing on a urine sample compared with vaginal self-collected or cervical (clinician-collected) samples
* To assess the efficacy of treatment in terms of post-treatment cervical lesions

Methodology. Participants will be WLHIV aged 25 to 49 and eligible for CC screening. Health care workers will also be invited to participate to the implementation research. The data collected will be quantitative and qualitative.

DETAILED DESCRIPTION:
Context. Cervical cancer (CC) is a leading cause of death among women living with HIV (WLHIV) in resource-limited settings. There is compelling evidence that screening for human papillomavirus (HPV) infection by testing is a very sensitive method for identifying women at risk for precancerous lesions of the cervix. But since HPV infections are very common among WLHIV, it is necessary to have secondary triage to identify women who need to be treated.

The HPV-based screening approach includes multiple steps, and dropout may occur at these different steps, compromising the success of the CC elimination strategy. A single-visit screen and treat approach has been recommanded based on the results of a large South African trial. Yet, in many contexts, including those with limited resources, the screening and treatment activities are often performed in multiple visites for logistical reasons, resulting in many dropouts. Strategies based on the differentiated prestation approach, which propose a simplified management centered on the patients preferences, could guide the adaptation of the single-visit approach to account for contextual constraints while maintaining high effectiveness.

The OptiTri-GC study aims to design and assess the impact of a differentiated CC screen and treat strategy in a district hospital; It will assess both its implementation and its effectiveness based on the completeness at each stage of the screening cascade. In addition, it will also include three sub-studies designed to evaluate :

* the performance of urinary HPV testing.
* the performance of different post-HPV test triage options (partial genotyping, simple or Artifical Intelligence assisted visual inspection, methylation markers)
* the risk of post-treatment cervical disease and the performance of different cure markers.

This will be a type 2 hybrid study that combines intervention research and implementation research. A quasi-experimental design ("before - after") combined with case study will be used for the effectiveness component of the research. During the first period, a single visit approach will be used while differentiated approach will be prepared using participatory research. During the second period, the differentiated approach will be implemented.

The general objective of this research is to assess the (cost-)effectiveness and implementation of different the two screening delivery strategies.

Main specific objectives include:

* To assess the effectiveness of each implementation strategy (in terms of cascade completeness)
* To assess the implementation of each strategy in terms of :

  * Success through the measure of fidelity, reach and completeness
  * Identification of adaptation, barriers and facilitating/leverage factors
  * Perception, feasibility and acceptability of the screening strategies (by patients and health care workers)
* To assess the participants' stress levels during the screening process and to identify potential psychosocial support strategies
* To document the experience of WLHIV and health workers during the screening process and the post-treatment follow-up.
* To assess the performance of different triage methods among HPV+ participants (partial genotyping, simple or aided visual inspection, S5 methylation)
* To assess the performance of HPV testing on a urine sample compared with vaginal self-collected or cervical (clinician-collected) samples
* To assess the efficacy of thermal ablation treatment in terms of post-treatment cervical lesions

Methodology. The implementation research will combine quantitative and qualitative methods and will be based on the i-PARHIS model. Participants will be WLHIV aged 25 to 49 and eligible for CC screening. Health care workers will also be invited to participate to the implementation research. The data collected will be quantitative and qualitative. Biomedical data will be collected prospectively. The implementation data will combine routine monitoring data, cross-sectional surveys, interviews and observations. The analysis will be sequential or convergent depending on the stages of the project.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* receiving antiretroviral therapy
* living in the department of the study hospital

Exclusion Criteria:

* ongoing pregnancy
* hysterectomy
* treatment of cervical lesion in the past 12 months
* Expected follow-up difficulties: planned absence that could interfere with the participation in the study (e.g., travel abroad, relocation, imminent transfer, etc.);
* Any pathology or concomitant treatment which, in the opinion of the investigators, contraindicates participation or prevents satisfactory participation in the study Inclusion deferred if
* menstrual bleeding
* post-partum (<12 weeks after delivery)
* clinicla signs of cervical or pelvic infection

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1422 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Screening completeness | 60 days post screening initiation
  Proportion of HPV+ participants completing all screening steps within 60 days of inclusion.

SECONDARY OUTCOMES:
Screening completeness 2 | 120 days post screening initiation
  Proportion of HPV+ participants completing all screening steps within 120 days of inclusion.
Acceptability of the screening delivery strategy | Baseline (screening)
  Questionnaire assessing the acceptability and using a 4 point Likert scale
Triage performance | Baseline (screening)
  Sensitivity, specificity of the triage option to detect CIN2+ and CIN3+ lesion
Performance of urinary HPV test | Baseline (screeening)
  Concordance between HPV test results from urine samples and those from cervical specimen collected by the clinician
Post treatment cervical lesion | 12 months
  Frequency of CIN2+ lesion 12 months after treatment and performance of the markers of cure (sensitivity and specificity)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Debeaudrap, MD, PhD, Study Director — Institut de Recherche pour le Développement (IRD); Joëlle Sobngwi, MD, PhD, Principal Investigator — RSD Institute
Locations (1):
- Foumban hospital, Foumban, Cameroon

IPD SHARING:
Plan to Share IPD: No